CLINICAL TRIAL: NCT04558346
Title: Ghrelin (OXE--103) for Acute Concussion Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Rippee (Other)
Collaborators: University of Kansas Health System (Other); University of Kansas Medical Center (Other)
Responsible Party: Sponsor-Investigator, Michael Rippee, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00145983
Record Dates: First submitted 2020-09-03; First posted 2020-09-22 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Concussion, Brain; Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic | interventions — Ghrelin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (40ug/kg) will be self-administered twice daily for 14 days.
  ONLY THE PART B (ACUTE) SUBJECTS WILL BE RANDOMIZED AND MAY RECEIVE PLACEBO.
  Interventions: Drug: Placebo
- Ghrelin (OXE-103) (Experimental): OXE-103 (40ug/kg) will be self-administered twice daily for 14 days.
  PART A (POST-ACUTE) SUBJECTS WILL BE OFFERED EXPERIMENTAL TREATMENT WITHOUT RANDOMIZATION.
  PART B (ACUTE) SUBJECTS WILL BE DOUBLE-BLIND RANDOMIZED TO EXPERIMENTAL OR PLACEBO TREATMENT.
  Interventions: Drug: Ghrelin (OXE-103)

INTERVENTIONS:
Drug: Ghrelin (OXE-103) — 40ug/kg twice daily by self-injection
  Arms: Ghrelin (OXE-103)
Drug: Placebo — 40ug/kg twice daily by self-injection
  Arms: Placebo

SUMMARY:
Concussions are the leading form of mild traumatic brain injury. Management of concussions and mild traumatic brain injury is a high priority medical focus, social concern, and research topic. Currently, there are no FDA approved treatments for acute concussion. The current standard of care is rest followed by gradual return to normal activity. The purpose of this study is to show improvement in the way patients feel or function after a concussion.

OXE-103 is a protein hormone produced in the laboratory which identical to the hormone ghrelin that is secreted by the stomach. This study will investigate the use of this hormone as treatment for symptoms of acute concussion. The goal of this study is to show improvement in the way study participants feel or function after concussion.

An OXE-103 (ghrelin) agonist is already FDA approved for another condition, but not for concussion. For concussion, it is considered investigational.

This study will examine, if ghrelin is taken every day for two weeks, if the brain will heal faster and help improve or resolve symptoms. The study will also include a placebo arm and a non-treatment group (for those who wish to participate but do not want to receive any treatment). The OXE-103 and placebo will be self-administered through injections using needles.

DETAILED DESCRIPTION:
All consenting participants will be screened for eligibility.

The study does not include randomization and all enrolling subjects will be offered treatment with OXE-103. Enrolling subjects will also have the option to choose participation in a non-treatment control group if they do not want treatment.

Consenting participants must be willing to commit to the following:

* give themselves subcutaneous injections twice a day (for the treatment groups)
* attend several study visits, which require both in-person and phone-only visits
* complete various questionnaires and testing
* have blood drawn
* have ECG's performed
* undergo a pregnancy test (if of childbearing potential) and use contraception while on study (for the treatment groups)
* tell the study team about any side effects they might experience from the study drug during study participation

Total participation will last about 7 weeks, which includes screening, 14 days of taking the study drug, and 4 weeks of follow-up. Participation for the non-treatment group will last the same amount of time.

ELIGIBILITY:
INCLUSION AND EXCLUSION:

Subjects must be consented within 28 days post injury.

Subjects will have a symptom severity score of at least 20 at the time of randomization in order to reduce the expected degree (number and severity) of spontaneous symptom resolution prior to study completion.

Subjects with pre-existing neurologic conditions other than mTBI (including cognitive dysfunction) will be excluded.

Subjects receiving, or planning to receive, a continuous ketamine infusion while enrolled in study will be excluded.

Subjects with these known endocrinological abnormalities at baseline will be excluded from study: diabetes mellitus, excess or deficiency of growth hormone, cortisol, or prolactin. Exclusion from study for any other endocrinological abnormalities or diagnoses existing at baseline are ultimately up to the discretion of the study physician.

Significant abnormalities in serum creatinine (>2.5 mg/dL), or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times the upper limit of normal, or bilirubin (>2.5 mg/dL) will exclude subjects from participation.

Subjects with any abnormal findings noted on imaging, such as hemorrhage, will be excluded from the study. Subjects who meet criteria for moderate or severe TBI will also be excluded.

Subjects who are known to be pregnant will be excluded. Subjects who do not agree to double-barrier contraception or abstinence (for female subjects of child-bearing potential or male subjects who are sexually active with a female of child-bearing potential) until the day following last dose (total of at least 5 half-lives) will be excluded.

Subjects receiving other concomitant medications, physical therapy, or other treatments related to their current mTBI will be eligible if they meet the inclusion criteria.

Subjects (or household members) who are not able to inject themselves or the subject will be excluded.

Subjects are not allowed to be concurrently enrolled in another therapeutic intervention clinical trial while participating in this study. Any subjects currently enrolled in such a separate therapeutic intervention clinical trial, for any condition, will be excluded from participating in this study. For clarification, this does not include observational clinical trials or registries.

Ultimately study subject participation will be at the discretion of the study physician.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rippee, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Standard of Care: Placebo (40ug/kg) will be self-administered twice daily for 14 days.
  ONLY THE PART B (ACUTE) SUBJECTS WILL BE RANDOMIZED AND MAY RECEIVE PLACEBO. PART A (POST-ACUTE) SUBJECTS WILL ONLY RECEIVE STANDARD OF CARE (PHYSICAL THERAPY, SYMPTOMATIC TREATMENTS)
  Placebo: 40ug/kg twice daily by self-injection
- Ghrelin (OXE-103): OXE-103 (40ug/kg) will be self-administered twice daily for 14 days.
  PART A (POST-ACUTE) SUBJECTS WILL BE OFFERED EXPERIMENTAL TREATMENT WITHOUT RANDOMIZATION.
  PART B (ACUTE) SUBJECTS WILL BE DOUBLE-BLIND RANDOMIZED TO EXPERIMENTAL OR PLACEBO TREATMENT.
  Ghrelin (OXE-103): 40ug/kg twice daily by self-injection
Period: Overall Study
Arm/Group | Placebo/Standard of Care | Ghrelin (OXE-103)
Started | 8 | 15
Completed | 6 | 13
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Standard of Care | Ghrelin (OXE-103) | Total
Number analyzed (Participants) | 8 | 15 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [30 to 43] | 42 [41 to 51] | 42 [35 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 14 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 15 | 23

OUTCOME MEASURES:

1. Primary Outcome: Symptom Management - Post Concussion Symptom Scale
Description: The primary goal is to describe the change in severity of symptoms in sub-acute concussion with treatment with OXE-103 using the Post Concussion Symptom Scale questionnaire during the intervention period at days 1 and 15 as well as during the post-treatment period at day 44.
  The Post Concussion Symptom Scale questionnaire consists of 23 common concussion symptoms which are assigned a ranking of severity on a scale from 0 (no symptom) to 6 (severe symptom). This tool is used to capture both severity of concussion symptoms as well as the number of symptoms. Data will be reported with the total values of all 23 subscale symptoms (total score = sum of all subscale symptom scores)--total can range from 0 to 138 with lower scores indicating lower symptom burden and higher scores a higher symptom burden (lower score = better outcome)
Time Frame: Days 1, 15, and 44
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Standard of Care: STANDARD OF CARE (PHYSICAL THERAPY, SYMPTOMATIC TREATMENTS)
- Ghrelin (OXE-103): Ghrelin (OXE-103): 40ug/kg will be self-administered twice daily for 14 days.
Arm/Group | Standard of Care | Ghrelin (OXE-103)
Number analyzed (Participants) | 6 | 13
score on a scale
  Day 1 | 44 [28 to 71] | 71 [47 to 73]
  Day 15 | 39 [28 to 68] | 51 [24 to 69]
  Day 44 | 45 [6 to 67] | 20 [7 to 43]
  Change Day 15-Day 1 | -1 [-14 to 4] | -21 [-30 to -6]
  Change Day 44-Day 1 | -7 [-22 to 16] | -34 [-44 to -24]

2. Secondary Outcome: Quality of Life - QOLIBRI-OS
Description: A secondary goal is to examine change in quality of life with treatment of sub-acute concussion using the Quality of Life after Brain Injury The QOLIBRI scores are reported on a 0-100 scale , where 0=worst possible quality of life and 100=best possible quality of life.
  Responses to the 'satisfaction' items (i.e. items on the Cognition, Self, Daily Life & Autonomy, and Social Relationships scales) are on a 1-5 scale, 1= "not at all satisfied" and 5="very satisfied". Responses to the 'bothered' items (i.e. items on the Emotions and Physical Problems scales) are reverse scored to correspond with the satisfaction items, where 1="very bothered" and 5="not at all bothered".
  The responses on each scale are summed to give a total, and then divided by the number of responses to give a scale mean. The scale means have a maximum possible range of 1 to 5. In a similar manner the QOLIBRI Total score is calculated by summing all the responses, and then dividing by the actual number of responses.
Time Frame: Days 1, 15, and 44
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Groups:
- Ghrelin (OXE-103): Ghrelin (OXE-103): 40ug/kg twice daily by self-injection for 14 days
Arm/Group | Standard of Care | Ghrelin (OXE-103)
Number analyzed (Participants) | 6 | 13
score on a scale
  Day 1 | 13 [11 to 14] | 8 [7 to 15]
  Day 15 | 11 [7 to 17] | 17 [8 to 19]
  Day 44 | 10 [7 to 18] | 18 [12 to 23]
  Change Day 15-Day 1 | 1 [-4 to 6] | 2 [1 to 6]
  Change Day 44-Day 1 | 1 [-6 to 5] | 5 [3 to 12]

ADVERSE EVENTS:
Time Frame: 44 days
Arm/Group | Placebo/Standard of Care | Ghrelin (OXE-103)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/15
Other Adverse Events (participants affected / at risk) | 0/6 | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Standard of Care (N=6) | Ghrelin (OXE-103) (N=15)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3
Injection site pain (Skin and subcutaneous tissue disorders) | 0 | 5
Nausea (Gastrointestinal disorders) | 0 | 4
Edema (Skin and subcutaneous tissue disorders) | 0 | 1 — Swollen foot
Diarrhea (Gastrointestinal disorders) | 0 | 2
Bruising (Skin and subcutaneous tissue disorders) | 0 | 8 — Bruising at injection site
Headache (Nervous system disorders) | 0 | 1
Gastroesophageal reflux (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 0 | 4
Infection (Infections and infestations) | 0 | 1 — COVID
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Hot flash (Vascular disorders) | 0 | 2
Stomach Gurgling (Gastrointestinal disorders) | 0 | 7
Insomnia (General disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 8
Dizziness (Nervous system disorders) | 0 | 2
Bloating (Gastrointestinal disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2
Vivid dreams (General disorders) | 0 | 1
Increased thirst (Metabolism and nutrition disorders) | 0 | 2
Increased ALT (Grade 2) (Investigations) | 0 | 1
Increased AST (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT04558346/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT04558346/SAP_001.pdf